CLINICAL TRIAL: NCT04638998
Title: Assessing Neuroinflammation in Gulf War Illness With Whole-Brain Magnetic Resonance Spectroscopy
Brief Title: Assessing Neuroinflammation in GWI Using MRS
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jarred Younger, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-3000004528; W81XWH-19-1-0725 (Other Grant/Funding Number: Department of Defense- Gulf War Illness Research Program)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Gulf War Syndrome
Keywords: neuroinflammation; Gulf War Illness
MeSH Terms: conditions — Persian Gulf Syndrome; Neuroinflammatory Diseases | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: The healthy control group are men ages 46-70 who were present in the Persian Gulf War between 1990 and August 1991. This cohort do not experience any Gulf War Illness symptoms.
  Interventions: Procedure: Magnetic Resonance Spectroscopic Imaging; Procedure: Blood draw
- Gulf War Illness: The GWI cohort are men ages 46-70 who were present in the Persian Gulf War between 1990 and August 1991. The men in this cohort will also meet the Kansas Inclusion Criteria for GWI.
  Interventions: Procedure: Magnetic Resonance Spectroscopic Imaging; Procedure: Blood draw

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopic Imaging — MRSI is a non invasive imaging technique used to detect neuroinflammation.
  Other Names: MRSI
Procedure: Blood draw — Blood will be drawn to assess systemic inflammation in Gulf War verterans.

SUMMARY:
The primary aim of this study is to determine if Gulf War Illness (GWI) likely involves neuroinflammation. The investigators hypothesize that GWI involves neuroinflammation. By assessing the five neuroinflammatory outcomes across the brain, the investigators can determine if there are focal or global signs of one or more neuroinflammatory markers in the brains of individuals with GWI. This neuroimaging technique may allow investigators and others to detect cases of GWI neuroinflammation, which would improve treatment decisions as well as the development of new targeted therapies. It is an ideal diagnostic tool because it has low patient risk, is noninvasive, can be used repeatedly in longitudinal studies, provides whole-brain coverage, yields multiple independent markers of inflammation, and can be employed at most hospitals and research neuroimaging suites.

DETAILED DESCRIPTION:
This proposal is for a Tier 1 (Discovery) study that uses a human, cross-sectional, observational neuroimaging approach to measure neuroinflammation in Gulf War Illness (GWI). A whole-brain magnetic resonance spectroscopic imaging (MRSI) scan will be used to detect multiple markers of neuroinflammation in 30 individuals with GWI and 30 healthy veteran controls. The investigators have fully tested the MRSI scan in several patient groups, and have found strong evidence of neuroinflammation in fibromyalgia and chronic fatigue syndrome - conditions the investigators believe involve abnormal central immune system processing. The investigators have not, however, performed the scan on individuals with GWI. The discovery study will allow investigators to transfer this existing technology to the GWI field. This project meets the core Special Interest of investigating dysregulation between the immune and neurological systems in the brain.

The investigators' central hypothesis is that GWI involves chronic neuroinflammation. The symptoms of GWI (e.g. fatigue, musculoskeletal pain, sleep disturbances, and cognitive dysfunction) overlap heavily with classic cytokine-induced sickness responses. In the case of GWI, microglial cells in the brain can be pushed into a hypersensitized state by toxins or abnormal immune challenges, leading to chronic overproduction of pro-inflammatory factors that result in the primary symptoms of GWI.

To test the central hypothesis, it is necessary to measure neuroinflammation in humans in vivo. However, most techniques are too invasive for use in living individuals. To address that problem, the investigators use an MRSI scan which provides metabolite concentrations in 4,000 separate voxels, giving whole-brain coverage. The scan yields measurements for: Myo-inositol (a marker of glial cell proliferation), lactate (a product of anaerobic metabolism), choline (a sign of cellular breakdown), and N-acetylaspartate (a marker of neuronal health). The scan also provides absolute brain temperature, which is shown to be elevated with severe neuroinflammation. The five main outcomes are as follows:

Myo-inositol (MI): Higher values represent greater microglia proliferation or gliosis.

Lactate (Lac): Higher values represent more severe inflammatory activity.

Choline (Cho): Higher values indicate greater cell turnover (inflammation, gliosis, or demyelination).

NAA: Lower values represent neurodegeneration.

Temperature: Higher values represent greater neuroinflammation. Metabolite and water-reference data will be analyzed using the MIDAS package and thermometry extension41. Absolute brain temperatures (in °C) within each voxel will be calculated by measuring the distance of the temperature-invariant NAA peak from the temperature-variant water peak using the formula: Tbrain = -102.76 × Δwater-NAA + 310.5°C, which has been validated in our scanner to produce reliable readings. Temperature will be expressed on absolute values in °C.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 46 and 70
* Veterans who meet the Kansas inclusion criteria .The Kansas Inclusion Criteria are a set of the most frequently reported symptoms experienced by Gulf War veterans. This frequency and severity of the symptoms reported by the participant indicate whether the person has Gulf War Illness or not. The Kansas Inclusion Criteria is the gold standard for identifying veterans with GWI in the field. The criteria are attached.
* Present in Persian Gulf between 1990 and August 1991
* Forward deployed (in Iraq or Kuwait)

Exclusion Criteria:

* Usage of experimental medications, opioid analgesics, psychostimulants (except caffeine), or benzodiazepines
* Uncontrolled diabetes, autoimmune disorders, and thyroid disorders.
* Major cardiovascular illness, cancer, or have any contraindications for MRI (including metallic implants or claustrophobia)

Ages: 46 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study requires the recruitment of Gulf War Veterans who were present in the Persian Gulf between 1990 and August 1991 and who were forward deployed to either Iraq or Kuwait. Of the approximate 650,000 service members who served in the Gulf War, only around 50,000 were women. As the number of female veterans who fit the study criteria wanes in comparison to that of the male veterans, it would prove extremely difficult to recruit both GWI and age-matched, healthy control female veterans. To circumvent this issue, the investigators chose to use only male Gulf War veterans for our study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Jones C, Haskin O, Younger J. Neurometabolite alterations in Gulf War Illness: a whole-brain magnetic resonance spectroscopy study. Exp Brain Res. 2025 Oct 25;243(11):237. doi: 10.1007/s00221-025-07174-w. PMID 41137912

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control | Gulf War Illness
Started | 21 | 28
Completed | 20 | 25
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Gulf War Illness | Total
Number analyzed (Participants) | 21 | 28 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 28 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 28 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 19 | 23 | 42
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 28 | 49

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Myoinositol in the Brain
Description: The concentration of myoinositol will be measured in the brain using MRI as a measure of neuroinflammation. This will be measured in both the control and experimental groups.
Time Frame: 20 minutes
Population: Some participants data were excluded due to poor quality
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Arm/Group | Healthy Control | Gulf War Illness
Number analyzed (Participants) | 19 | 20
Institutional Units (IU) | 0.001260 (0.0002362) | 0.001205 (0.0001699)

2. Primary Outcome: Concentration of Lactate in the Brain
Description: The concentration of lactate will be measured in the brain using MRI as a measure of neuroinflammation. The concentration will be expressed in water-normed "Institutional Units". This will be measured in both the control and experimental groups. Values are expressed as metabolites averaged across the cortical lobes and cerebellum.
Time Frame: 20 minutes
Population: Some participants data were excluded due to poor quality
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Arm/Group | Healthy Control | Gulf War Illness
Number analyzed (Participants) | 19 | 20
Institutional Units (IU) | 0.0003886 (0.0001629) | 0.0005388 (0.000365)

3. Primary Outcome: Concentration of Choline in the Brain
Description: The concentration of choline will be measured in the brain using MRI as a measure of neuroinflammation. This will be measured in both the control and experimental groups.
Time Frame: 20 minutes
Population: Some participants data were excluded due to poor quality
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Arm/Group | Healthy Control | Gulf War Illness
Number analyzed (Participants) | 19 | 20
Institutional Units (IU) | 0.0003838 (0.000051446) | 0.0003499 (0.000034982)

4. Primary Outcome: Concentration of N-acetylaspartate in the Brain
Description: The concentration of N-acetylaspartate will be measured in the brain using MRI as a measure of neuroinflammation. This will be measured in both the control and experimental groups.
Time Frame: 20 minutes
Population: Some participants data were excluded due to poor quality
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Arm/Group | Healthy Control | Gulf War Illness
Number analyzed (Participants) | 19 | 20
Institutional Units (IU) | 0.0023191 (0.0001821) | 0.0022186 (0.0001721)

5. Primary Outcome: Temperature in the Brain
Description: The temperature of the brain will be measured using MRI as a measure of neuroinflammation. This will be measured in both the control and experimental groups. An amplitude-weighted combination of NAA, creatine, and choline was used as the reference for temperature deviations.
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Healthy Control | Gulf War Illness
Number analyzed (Participants) | 19 | 20
degrees Celsius | 36.622 (0.322) | 36.826 (0.331)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Healthy Control | Gulf War Illness
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/28
Other Adverse Events (participants affected / at risk) | 0/21 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04638998/Prot_SAP_000.pdf